CLINICAL TRIAL: NCT00111241
Title: Assessment of Knee Joint Articular Cartilage Volume Change, Bone Loss and Change in Body Composition in Women Treated With Anastrozole or Letrozole and Comparison With Untreated Controls
Brief Title: Changes in Knee Articular Cartilage Volume in Women on Aromatase Inhibitors
Status: Completed | Type: Observational
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Professor Susan Davis, Professor of Women's Health, Monash University
Other Study IDs: 2004/949
Record Dates: First submitted 2005-05-18; First posted 2005-05-19 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-11

CONDITIONS: Arthralgia
Keywords: bone fracture; cartilage; osteoporosis; breast cancer; aromatase inhibitors; knee articular cartilage volume
MeSH Terms: conditions — Arthralgia; Fractures, Bone; Osteoporosis; Breast Neoplasms | interventions — Aromatase Inhibitors; Letrozole; Anastrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: aromatase inhibitors (letrozole, anastrozole) — Women prescribed an aromatase inhibitor by their clinician were compared with healthy controls in the community who had been recruited to a prior study
  Other Names: no other names

SUMMARY:
Many women with breast cancer are treated with a class of drugs called aromatase inhibitors (mainly letrozole or anastrozole), which lowers the amount of estrogen being produced in the body. Women on aromatase inhibitors appear to experience joint pains and arthralgia. The aim of this study is to determine whether the joint pains experienced by some women on aromatase inhibitors is associated with more defects in their cartilage, compared to women not receiving this therapy. Using the magnetic resonance imaging (MRI) technique, the knee joint will be examined to assess changes in cartilage volume over time.

DETAILED DESCRIPTION:
The mechanism of increased bone loss and fracture risk is clearly related to the depletion of estrogen production in the bone. But why there is a higher rate of reporting arthralgia, fracture and joint pain amongst women on aromatase inhibitors is not understood.

Using magnetic resonance imaging (MRI) to measure knee articular cartilage volume, we have demonstrated that post menopausal hormone therapy used for at least five years is associated with retention of articular cartilage in the knee, indicating that oestrogen may protect against the development of osteoarthritis in post menopausal women. Furthermore, we have recently observed that free testosterone is associated with loss of tibial cartilage, after taking into account age, body mass index, baseline tibial cartilage volume, tibial plateau area and total bone mineral content in healthy men. Whether an excess of testosterone to oestrogen as a consequence of aromatase inhibition has an adverse effect on articular cartilage volume warrants further investigation.

This study will include non-hysterectomised women aged 40 to 65 years who have undergone breast surgery and then commenced on aromatase inhibitors within the preceding 12 weeks. The control group (which has been fully recruited) included non-hysterectomised, healthy women aged 40 to 65 years. A MRI of the dominant knee will be used to compare changes in knee articular volume over time. A MRI will be done at baseline and again at 2 years. Changes in knee articular volume is the primary outcome. We will also use this opportunity to compare menopausal symptoms (assessed using the Menopause Quality of Life (MENQOL)questionnaire) between women treated with aromatase inhibitors and those who are not. Well-being will also be assessed using the Psychological General Well-Being index.

ELIGIBILITY:
Inclusion Criteria:

Group 1 :

* Aged 40 - 65
* Non-hysterectomised women who have undergone breast surgery
* Women on aromatase inhibitors within preceding 12 weeks

Group 2 : control group

* Healthy, non-hysterectomised women aged 40-65 .

Exclusion Criteria:

* Previous knee injury requiring non-weight bearing treatment for > 24 hrs or surgery (including arthroscopy)
* Inability to complete the study (eg proposed relocation)
* Contraindication to undergoing an MRI including pacemaker, metal sutures, presence of shrapnel, iron filings in eye
* Claustrophobia

Additional Exclusions for Group 1

* Treatment with tamoxifen for > 8 weeks prior to commencement
* Knee pain lasting for >24 hours in the last 5 years (prior to commencement on anastrozole or letrozole)
* Anastrazole or Letrozole therapy for > 12 weeks

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be informed of study by their treating physician and invited to participate and by community sample.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2005-05; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Davis, MBBS PhD, Principal Investigator — Director Women's Health Program
Locations (1):
- Women's Health Research Program, Monash University, The Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Women With Breast Cancer: women with hormone receptor positive ( HR+) breast cancer, prescribed an aromatase inhibitor (AI)
- Healthy Control Group: healthy postmenopausal aged-matched controls from prior data base
Period: Overall Study
Arm/Group | Women With Breast Cancer | Healthy Control Group
Started | 45 | 70
Completed | 30 | 62
Not Completed | 15 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Protocol Violation | 9 | 8
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Women With Breast Cancer on Aromatase Inhibitor Therapy: women with hormone receptor positive breast cancer prescribed an aromatase inhibitor
- Control: healthy postmenopausal aged-matched controls from prior data base
- Total: Total of all reporting groups
Arm/Group | Women With Breast Cancer on Aromatase Inhibitor Therapy | Control | Total
Number analyzed (Participants) | 45 | 70 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 70 | 115
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 70 | 115
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 45 | 70 | 115

OUTCOME MEASURES:

1. Primary Outcome: Knee Cartilage Volume
Description: change in medial and lateral articular tibial cartilage volume over two years
Time Frame: Baseline, two years
Measure: Mean (Standard Deviation); unit: mm³
Groups:
- Women With Breast Cancer: women recruited with HR+ breast cancer prescribed an AI
Arm/Group | Women With Breast Cancer | Control
Number analyzed (Participants) | 30 | 62
mm³ | 2042 (151) | 1971 (207)

2. Secondary Outcome: Knee Subchondral Bone Expansion
Description: change in subchondral bone expansion area over two years
Time Frame: Baseline, Two years
Measure: Mean (Standard Deviation); unit: mm²
Groups:
- Healthy Control Group: postmenopausal, nonhysterectomized, women not taking hormone replacement therapy,and with a body mass(BMI) between 20 and 37 kilograms per metre squared (kg/m2)
Arm/Group | Women With Breast Cancer | Healthy Control Group
Number analyzed (Participants) | 45 | 70
mm² | 2020 (180) | 1992 (204)

ADVERSE EVENTS:
Time Frame: Baseline, 2 years
Groups:
- Women With Breast Cancer: Of 45 women recruited with HR+ breast cancer prescribed an AI, 30 women provided paired MRI data, including 1 woman who withdrew at 0.8years due to metastatic disease. 3 women did not have even a baseline MRI (2 gave no reason and one withdrew with joint pain), 2 had no follow-up MRI, one stopped her AI, 3 cited personal reasons, one withdrew due to cancer complications, 3 changed to tamoxifen, one was lost to follow up and one gave no reason for withdrawal.
- Control Group: Of 70 women participating as controls, 8 had missing MRI data
Arm/Group | Women With Breast Cancer | Control Group
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/70
Other Adverse Events (participants affected / at risk) | 0/45 | 0/70

LIMITATIONS AND CAVEATS:
Menopausal Symptoms and Well-being were previously entered as Secondary Outcome Measures. Data not available to assess these outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes